CLINICAL TRIAL: NCT05232149
Title: A Randomized, Multi-center, Adaptive Phase IIa/IIb Study to Evaluate the Efficacy and Safety of Orelabrutinib in Adult Patients With Persistent or Chronic Primary Immune Thrombocytopenia
Brief Title: A Study to Evaluate the Efficacy and Safety of Orelabrutinib in Adult Patients With Immune Thrombocytopenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-00116
Record Dates: First submitted 2021-12-20; First posted 2022-02-09 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Primary Immune Thrombocytopenia
Keywords: Persistent or chronic
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Bronchiolitis Obliterans Syndrome | interventions — orelabrutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lower Dose (Experimental): Orelabrutinib is a white, round, uncoated tablet
  Interventions: Drug: Orelabrutinib( lower dose)
- Higher Dose (Experimental): Orelabrutinib is a white, round, uncoated tablet
  Interventions: Drug: Orelabrutinib( higher dose)

INTERVENTIONS:
Drug: Orelabrutinib( lower dose) — Orelabrutinib is a white, round, uncoated tablet, will be taken lower dose QD by patients with persistent or chronic primary immune thrombocytopenia
  Arms: Lower Dose
Drug: Orelabrutinib( higher dose) — Orelabrutinib is a white, round, uncoated tablet, will be taken higher dose QD by patients with persistent or chronic primary immune thrombocytopenia
  Arms: Higher Dose

SUMMARY:
The study is designed to be a randomized, open, multi-center, phase IIa/IIb seamless adaptive trial.

Phase IIa: The study consists of a screening period, a core treatment period, an open label extension period, and a safety follow-up period Phase IIb: At present, a preliminary exploratory study (i.e., phase IIa study) will be conducted first. The design of the phase IIb study (including the selection of populations) will be clarified after a relatively clear understanding of the therapeutic effect, value, risks and benefits of the BTK inhibitor for ITP is obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects have had a detailed understanding of the nature, significance, possible benefits, possible inconveniences, and potential risks of the trial, understood the study procedures, and voluntarily signed a written ICF before the study.
2. Males or females aged from 18 to 80 years (including the marginal values).
3. With a body weight of ≥ 35 kg at screening.
4. Diagnostic criteria:the diagnosis of persistent (3-12 months) or chronic (≥ 12 months) ITP is met
5. Patients who have failed at least 1 prior first-line standard therapy for ITP, or who have failed to tolerate a standard therapy.
6. Women of childbearing potential must take a complementary barrier method of contraception in combination with a highly effective method of contraception at screening, throughout the trial, and within 90 days after the last dose of the investigational drug.
7. The mean of two platelet counts is less than 30 × 109/L and no platelet count is greater than 35 × 109/L during the screening visit and/or before the first dose.

Exclusion Criteria:

1. Severe hemorrhage occurred within 4 weeks prior to screening.
2. Subjects suffer from severe ITP at screening
3. Subjects have other diseases which mention in protocol
4. Subjects develop intracranial hemorrhage within 6 months prior to screening.
5. Active and uncontrollable infection
6. Subjects have a history of coagulopathy other than ITP
7. Subjects with a history of malignancies.
8. History of major organ transplantation or hematopoietic stem cell/bone marrow transplantation.
9. Subjects with a known history of hypersensitivity to the investigational drug as described in the Protocol, or any ingredients.
10. Subjects with a Medication history and surgical history which mention in protocol
11. Subjects do not meet the criterion of the laboratory test in protocol

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-21 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with the platelet count of ≥ 50 × 109/L after 12 weeks of treatment | 12 weeks

SECONDARY OUTCOMES:
Proportion of subjects who achieve a complete response (CR) over treatment time. CR is defined as a post-treatment platelet count of ≥100 × 109/L | 25 weeks
Occurrence of treatment emergent adverse events (TEAE) and treatment-related adverse events (TRAE) were evaluated according to severity | 25 weeks

OTHER OUTCOMES:
Cmax | 25 weeks
  To obtain pharmacokinetic (PK) data of Orelabrutinib include the peak plasma concentration (Cmax)

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Hainan People's Hospital, Haikou, Hainan
  - Henan Tumor Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - First Hospital of Nanchang University, Nanchang, Jiangxi
  - QiLu Hospital of Shandong University, Jinan, Shandong

REFERENCES:
- [Derived] Yan S, Zhou H, Huang R, Wang F, Mei H, Lin L, Guo J, Zhou X, Li Z, Liu Y, Li S, Zhou W, Hou Y, Hou M. A phase 2 trial of orelabrutinib showing promising efficacy and safety in patients with persistent or chronic primary immune thrombocytopenia. Am J Hematol. 2024 Jul;99(7):1392-1395. doi: 10.1002/ajh.27303. Epub 2024 Mar 28. No abstract available. PMID 38546375